CLINICAL TRIAL: NCT04609657
Title: Liking Adaptation to Beverages With Varying Sweetness Levels After Prolonged Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2002
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Sweetness Liking Adaptation
Keywords: sweetness; liking; adaptation; intensity; low calorie sweetener; full sugar; carbonated soft drink; sensory; taste; dietary compensation; beverage; perception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Same packaging for all (cans). Color and flavor matched.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control beverage for Habitual full-calorie CSD cohort, n=28 (Placebo Comparator): Full sweetness (sugar) for 6 months
  Interventions: Other: Flavored carbonated soft drink (CSD)
- Control beverage for Habitual low-calorie CSD cohort, n=28 (Placebo Comparator): Full sweetness low calorie sweetener (LCS) with sweetness level matched to the full sweetness sugar control for 6 months
  Interventions: Other: Flavored carbonated soft drink (CSD)
- Test beverage 1 for Habitual full-calorie CSD cohort, n=28 (Active Comparator): Reduced sweetness (moderate sugar level) for 6 months
  Interventions: Other: Flavored carbonated soft drink (CSD)
- Test beverage 1 for Habitual low-calorie CSD cohort, n=28 (Active Comparator): Reduced sweetness low calorie sweetener (LCS) with sweetness level matched to the moderate sugar sweetness level for 6 months
  Interventions: Other: Flavored carbonated soft drink (CSD)
- Test beverage 2 for Habitual full-calorie CSD cohort, n=28 (Active Comparator): Step-wise sweetness reduction over 6 months. Month 1 is the full sweetness sugar control, followed by monthly sweetness reduction. Remains at the reduced sweetness level (moderate sugar level) from months 4-6.
  Interventions: Other: Flavored carbonated soft drink (CSD)
- Test beverage 2 for Habitual low-calorie CSD cohort, n=28 (Active Comparator): Step-wise sweetness reduction over 6 months. Month 1 is the low calorie sweetener (LCS) sweetness equivalent of the full sweetness sugar control, followed by monthly LCS sweetness reduction (reductions equivalent to the corresponding sugar reduction arm sweetness levels). Remains at the reduced sweetness level (LCS equivalent of moderate sugar sweetness level) from months 4-6.
  Interventions: Other: Flavored carbonated soft drink (CSD)

INTERVENTIONS:
Other: Flavored carbonated soft drink (CSD) — Beverage

SUMMARY:
This is a double-blind, controlled, parallel, randomized sensory study. The study will consist of two cohorts; habitual regular full-calorie Carbonated Soft Drink (CSD) consumers and habitual low-calorie CSD consumers. Each cohort will be randomized to one of 3 interventions for six months (24 weeks):

* Intervention 1: Control (full sweetness) beverage
* Intervention 2: Step-wise sweetness reduction series of beverages
* Intervention 3: Moderate sweetness (reduced sweetness) beverage

The primary outcome is to assess the perception changes in sweetness (magnitude scale) and sweetness liking (Likert scale) of a test product and a control product over a period of six months. The study endeavors to explore whether consumers of sweetened carbonated beverages can adapt liking to lower sweetness beverages after prolonged exposure of daily consumption of beverages with step-wise reduction of sweetness, or maintenance at reduced (moderate) sweetness.

Additional analysis will be to assess dietary compensation for sweetness in the step-wise and moderate reduction arms compared to the control arms (the full calorie and low calorie control beverages). Dietary analysis of calories and intakes of total sugar, added sugar, and servings of low-/non-calorie sweeteners will be assessed using a 3-day diet record pre-intervention and monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 25-55 years of age
2. Habitually consume regular or diet CSD
3. Willing and able to consume at least one orange CSD beverage daily for a total of 6 months and abstain from other sweetened beverages
4. Willing and able to complete questionnaires regarding dietary intake and sensory perception
5. Has internet access via computer, phone or other device and is able to maintain internet access throughout the trial in order to complete daily online questionnaires
6. Participant is judged to be in good health based on a verbal health query and the general health and lifestyle questionnaire
7. Participant is willing to maintain his or her habitual diet, smoking habits and physical activity patterns, including habitual use of study approved medications and/or dietary supplements throughout the study period
8. Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators

Exclusion Criteria:

1. Regular smoker (more than 1 cigarette per week)
2. History or presence of type 1 or 2 diabetes mellitus
3. Extreme dietary habits, including but not limited to vegetarian diets and intentional consumption of a high fiber diet, gluten-free, low-carb, vegan, ketogenic, and intermittent fasting (defined as intentional fasting for longer than 16 hours or alternate day fasting)
4. Extreme changes to physical activity
5. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period
6. Recent history (within 12 months of screening; Visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits)
7. Individual has a condition the Clinical Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the participant at undue risk
8. Dislike of citrus flavored CSDs
9. Participation in another clinical trial within past 30 days
10. People who have phenylketonuria (low calorie sweetened beverages contain aspartame)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Sweetness liking | Changes over a period of 6 months, measured at monthly intervals from month 0 (baseline) to month 6
  Likert Scale, 9 point scale from 1=Dislike extremely to 9=Like extremely
Sweetness intensity perception | Changes over a period of 6 months, measured at monthly intervals from month 0 (baseline) to month 6
  Magnitude scale ranging from Barely perceptible to Strongest imaginable sweetness

OTHER OUTCOMES:
Dietary compensation for sweetness | Changes over a period of 6 months, measured at monthly intervals from month 0 (baseline) to month 6
  3-day diet record to assess calories and intake of total sugar, added sugar, low-/non calorie sweeteners

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- BioFortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mah E, Kamil A, Blonquist TM, Rehm CD, Qu S, Stern P, Wilson AR. Change in liking following reduction in sweetness level of carbonated beverages: a randomized controlled parallel trial. Sci Rep. 2024 Nov 5;14(1):26742. doi: 10.1038/s41598-024-77529-w. PMID 39500957